CLINICAL TRIAL: NCT01382043
Title: Angiographic and IVUS Follow-up After Simultaneously Implanted Different Drug-eluting Stents in Same Individuals (AIFSIDDES)
Status: Completed | Type: Observational
Sponsor: Liuhuaqiao Hospital (Other)
Responsible Party: Liujian, Liuhuaqiao Hospital
Other Study IDs: LHQ09-002
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2011-06

CONDITIONS: Percutaneous Coronary Angioplasty
Keywords: percutaneous coronary angioplasty; zotarolimus-eluting stent; sirolimus-eluting stent; biodegradable polymer; biocompatible polymer

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endeavor Segment group
- Excel Segment Group

SUMMARY:
The safety and efficacy of drug-eluting stents (DES) with a biocompatible polymer have been demonstrated in randomized clinical trials as well as in real world practice. Theoretically, a new DES with a biodegradable polymer should reduce the incidence of late in-stent thrombosis, however, the long-term safety and efficacy of these stents remains unknown. This study was aimed to compare the safety and efficacy of the Excel DES with a biodegradable polymer to the Endeavor DES with a biocompatible polymer in same individuals.

ELIGIBILITY:
Inclusion Criteria:

* simultaneous implantation of one or more Endeavor stents and one or more Excel stents during the same index procedure
* willing to be followed up with coronary angiography and intravascular ultrasound at least one year post-procedure.

Exclusion Criteria:

* Patients were excluded from the study if they had more than two kinds of stents implanted or if the two study stents were implanted during separate interventional procedures or in coronary artery bridge vessel or restenotic lesions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patiemts who underwent simultaneous implantation of one or more Endeavor stents and one or more Excel stents during the same index procedure and were evaluated with coronary angiography and intravascular ultrasound (IVUS) at least one year post-procedure.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dingcheng Xiang, Dr., Principal Investigator — Liuhuaqiao Hospital
Locations (1):
- Liuhuaqiao Hospital, Guangzhou, GD, China